CLINICAL TRIAL: NCT04565613
Title: Protein Supplementation Versus Standard Feeds in Underweight Critically Ill Children: A Dual-Centre Randomized Controlled Pilot Trial
Brief Title: Protein Supplementation vs Standard Feeds in Underweight Critically Ill Children: A Dual-Centre Pilot RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Duke-NUS Graduate Medical School (Other); Singapore Clinical Research Institute (Other); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Jan Hau Lee, Senior Consultant, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/2742
Record Dates: First submitted 2020-09-15; First posted 2020-09-25 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Critically Ill
Keywords: Critically ill; Protein supplementation; Nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to enteral protein supplementation or standard care (no enteral protein supplementation) in a 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care group (No Intervention): The participants will receive feeding as per standard of care (without protein or any other supplementations).
- Study interventional group (Experimental): The participants will receive protein supplementation to reach a final goal of 1.5 g/kg/day of protein on full feeds.
  Interventions: Dietary Supplement: Enteral protein supplementation

INTERVENTIONS:
Dietary Supplement: Enteral protein supplementation — The participants in the study interventional group will receive protein supplementation to reach a final goal of 1.5 g/kg/day of protein on full feeds. This will be via 100% whey protein isolate (Nestle Beneprotein). Doses will be calculated on the patient's admission weight and rounded up to the nearest 1g. Doses will not be adjusted to account for weight changes in the PICU.
  Protein supplementation will continue for a total of 7 days from the start of enrolment into the study or until PICU discharge, whichever is earlier. If the patient is able to take solid feeds during the study intervention period, the intervention will be stopped. However, if the device required for feeding is removed but the patient takes milk/liquid feeds fully, protein supplementation will continue.
  Other Names: Protein isolate (Nestle Beneprotein)
  Arms: Study interventional group

SUMMARY:
This pilot trial is part of a long-term research program leading to a large trial to determine if a strategy of supplementing protein in a subset of critically ill children is superior to standard enteral nutrition care. The investigators hypothesize that protein supplementation to critically ill children with body mass index (BMI) z-score <0 reduces the length of stay in the paediatric intensive care unit (PICU) and hospital, as well as the duration of mechanical ventilation (MV).

DETAILED DESCRIPTION:
Protein malnutrition is prevalent among critically ill children and associated with poor clinical outcomes. Current guidelines for provision of protein in daily management of critically ill children in pediatric intensive care units (PICUs) are based on limited and not high-quality evidence. The current protein supplementation approach, "one-size-fits-all" nutrition prescription, may not be appropriate for every critically ill child. Given the heterogeneity of the patients admitted to the PICU, a targeted approach based on individuals' needs represents a potential advancement in PICU care.

The central hypothesis is that protein supplementation in PICU care leads to improved clinical outcomes in subgroups of patients only. The investigators propose a dual-centre pilot randomized controlled trial in Singapore with two major aims:

1. To obtain key information for planning and conducting a large-scale multicentre study in Asia; and
2. to evaluate the benefit of protein supplementation to critically ill children with body mass index (BMI) z-scores on PICU <0

The main clinical outcome of interest is total number of days of hospital stay (from PICU admission to hospital discharge). Two protein supplementation regimes (≥ 1.5g/kg/day vs. standard care) will be randomly allocated to PICU patients with body mass index (BMI) z-scores <0. The investigators will determine the effect of protein supplementation on total length of hospital stay and other clinical outcomes, and assess the impact of protein supplementation on acquired functional impairment of PICU survivors 6 months after hospital discharge. In addition, the investigators will explore whether muscle ultrasound is a biomarker for protein balance in pediatric critical illness.

Upon completion of this study, the investigators will have strong preliminary data to plan, refine their study approach, and execute a future large multi-centre study across Asia. These data will ultimately guide protein provision and nutritional management of patients in PICU setting.

ELIGIBILITY:
Inclusion Criteria:

1. Between 28 days and 18 years of age
2. Have a BMI z-score < 0 on PICU admission
3. Requires respiratory support in the form of invasive or non-invasive mechanical ventilation (CPAP or BiPAP) within 24-48 hours of PICU admission, and the attending physician expects the child to require any respiratory support for at least 48 hours of PICU admission
4. Requires enteral nutrition support for feeding (e.g., oro-gastric, nasogastric, gastrostomy, naso-jejunal, oro-jejunal)
5. Have an expected PICU stay of > 48 hours

Exclusion Criteria:

1. Are not expected to survive this PICU admission because of palliative care (e.g., do-not-resuscitate status) or limited life support
2. Progressive neuromuscular disease (e.g., spinal muscular atrophy, Duchenne or other muscular dystrophy, multiple sclerosis, amyotrophic lateral sclerosis)
3. Medical conditions where increased or decreased protein intake is required, including acute kidney injury (stage 3 KDIGO criteria), chronic kidney disease (stage 4 and 5), inborn errors of metabolism, fulminant liver failure, severe burn injury
4. Contraindications to enteral nutrition (e.g., gut hemorrhage, post-gastrointestinal surgery etc.)
5. Diagnosed cow's milk protein allergy
6. Parenteral nutrition
7. Premature infants who are less than corrected gestational age of 44 weeks (gestational age + weeks after birth)
8. Were previously enrolled in this trial
9. Are currently enrolled in a potentially confounding trial
10. Diagnosis of anorexia nervosa and other eating disorders
11. On extra-corporeal membrane oxygenation (ECMO) support
12. Conditions that required significant fluid restriction (≤75% of maintenance fluid) (e.g., post cardiac surgery etc.)

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible patients approached for consent | Throughout study period, over 36 months
  Number of eligible patients who are approached for consent
Proportion of participants receiving their first protein supplementation within 72 hours of enrolment | Throughout the study, over 24 months
  Number of patients who received protein supplementation within 72 hours of enrolment
Participant accrual rate | Throughout the study, over 24 months
  Average monthly enrolment at each centre
Protocol adherence | Throughout study period, over 24 months
  >80% of protein target administered according to the protocol in the intervention arm

SECONDARY OUTCOMES:
PICU mortality | Throughout study period, over 36 months
  Death in PICU
PICU length of stay | Throughout study period, over 36 months
  Duration of stay in the PICU
Hospital length of stay | Throughout the study period, over 36 months
  Duration of stay in the hospital
Adverse events | Throughout study period, over 36 months
  Development of adverse events such as feeding intolerance, diarrhoea, gastrointestinal bleeding
Change in muscle size | During PICU stay, PICU discharge, hospital discharge and 6 months follow-up
  Longitudinal change in muscle size as assessed by ultrasound. Muscles for assessment include rectus femoris and diaphragm
Anthropometry | During PICU stay, PICU discharge, hospital discharge and 6 months follow-up
  Change in anthropometric measurements
Functional status | PICU admission, hospital discharge and 6 months follow-up
  Assessment of functional status via functional status scale (FSS). FSS scores ranged from 6 to 30. A higher score denotes worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hau Lee, Principal Investigator — KK Women's and Children's Hospital, SingHealth
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Data from this pilot study may be used for the larger study. If so, these data will not be made available to other researchers till the larger study is completed or deemed not feasible.

REFERENCES:
- [Derived] Wong JJM, Ong JSM, Ong C, Allen JC, Gandhi M, Fan L, Taylor R, Lim JKB, Poh PF, Chiou FK, Lee JH. Protein supplementation versus standard feeds in underweight critically ill children: a pilot dual-centre randomised controlled trial protocol. BMJ Open. 2022 Jan 4;12(1):e047907. doi: 10.1136/bmjopen-2020-047907. PMID 34983751